CLINICAL TRIAL: NCT06679998
Title: A Dose-increasing, Randomized, Double-blind, Placebo-controlled, Single-dose/multiple-dose Phase I Clinical Trial Evaluating the Safety, Tolerability and Pharmacokinetics of AAPB for Injection in Healthy Chinese Subjects.
Brief Title: A Phase I Clinical Trial Evaluating the Safety, Tolerability and Pharmacokinetics of AAPB for Injection
Acronym: AAPB
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAPB-Ⅰ-KY001
Record Dates: First submitted 2024-11-04; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Acute Ischemic Stroke (AIS)
MeSH Terms: conditions — Ischemic Stroke | interventions — Infusions, Intravenous; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (14):
- Single administration of-AAPB-10mg group (Experimental): 10mg of AAPB for injection was administered as a single intravenous drip
  Interventions: Drug: Single dose, AAPB by injection, intravenous drip.
- Single dose - placebo -10mg group (Placebo Comparator): 10mg of placebo was administered as a single intravenous infusion
  Interventions: Other: Single dose, placebo, intravenous drip.
- Single administration of -AAPB-25mg group (Experimental): 25mg AAPB for injection.The drug was administered as a single intravenous drip
  Interventions: Drug: Single dose, AAPB by injection, intravenous drip.
- Single dose - placebo -25mg group (Placebo Comparator): 25mg of placebo was administered as a single intravenous infusion
  Interventions: Other: Single dose, placebo, intravenous drip.
- Single administration of -AAPB-50mg group (Experimental): 50mg AAPB for injection.The drug was administered as a single intravenous drip
  Interventions: Drug: Single dose, AAPB by injection, intravenous drip.
- Single dose - placebo -50mg group (Placebo Comparator): 50mg of placebo was administered as a single intravenous infusion
  Interventions: Other: Single dose, placebo, intravenous drip.
- Single administration of -AAPB-75mg group (Experimental): 75mg AAPB for injection.The drug was administered as a single intravenous drip
  Interventions: Drug: Single dose, AAPB by injection, intravenous drip.
- Single dose - placebo -75mg group (Placebo Comparator): 75mg of placebo was administered as a single intravenous infusion
  Interventions: Other: Single dose, placebo, intravenous drip.
- Single administration of-AAPB-100mg group (Experimental): 100mg AAPB for injection.The drug was administered as a single intravenous drip
  Interventions: Drug: Single dose, AAPB by injection, intravenous drip.
- Single dose - placebo -100mg group (Placebo Comparator): 100mg of placebo was administered as a single intravenous infusion
  Interventions: Other: Single dose, placebo, intravenous drip.
- Multiple administration-AAPB-A group for injection (Experimental): AAPB-A group dose for injection An intravenous drip. Once a day for 7 days
  Interventions: Drug: Multiple dosing, AAPB for injection, intravenous drip
- Multiple dosing -Placebo-A group (Placebo Comparator): Placebo, Group A dose, Intravenous infusion, Once a day for 7 days
  Interventions: Other: Multiple dosing, placebo, IV drip
- Multiple administration-AAPB-B group for injection (Experimental): AAPB-B group dose for injection An intravenous drip. Once a day for 7 days
  Interventions: Drug: Multiple dosing, AAPB for injection, intravenous drip
- Multiple dosing -Placebo-B group (Placebo Comparator): Placebo, Group B dose, Intravenous infusion, Once a day for 7 days
  Interventions: Other: Multiple dosing, placebo, IV drip

INTERVENTIONS:
Drug: Single dose, AAPB by injection, intravenous drip. — Subjects received a single intravenous infusion of AAPB for injection. Each dose of AAPB for injection was dissolved with 0.9% sodium chloride injection, the infusion volume was 100mL, once a day, and each time was continuously injected for 60 min±5min.
  Arms: Single administration of -AAPB-25mg group; Single administration of -AAPB-50mg group; Single administration of -AAPB-75mg group; Single administration of-AAPB-100mg group; Single administration of-AAPB-10mg group
Other: Single dose, placebo, intravenous drip. — Subjects received a single intravenous infusion of placebo. Each dose of placebo was dissolved by 0.9% sodium chloride injection with an infusion volume of 100mL once a day for 60 min±5min each time.
  Arms: Single dose - placebo -100mg group; Single dose - placebo -10mg group; Single dose - placebo -25mg group; Single dose - placebo -50mg group; Single dose - placebo -75mg group
Drug: Multiple dosing, AAPB for injection, intravenous drip — Subjects received AAPB for injection with multiple intravenous drips. Each dose of AAPB for injection was dissolved with 0.9% sodium chloride injection, the infusion volume was 100mL, once a day, 60 min±5min each time, for 7 consecutive days.
  Arms: Multiple administration-AAPB-A group for injection; Multiple administration-AAPB-B group for injection
Other: Multiple dosing, placebo, IV drip — Subjects received multiple intravenous doses of placebo. Each dose of placebo was dissolved by 0.9% sodium chloride injection with an infusion volume of 100mL once a day for 60 min±5min each time for 7 consecutive days.
  Arms: Multiple dosing -Placebo-A group; Multiple dosing -Placebo-B group

SUMMARY:
This is a Phase I clinical to evaluate the safety and tolerability of single and multiple intravenous infusions of AAPB at different doses over 7 consecutive days.

DETAILED DESCRIPTION:
This is a dose-increasing, randomized, double-blind, placebo-controlled, single-dose/multiple-dose phase I clinical trial evaluating the safety, tolerability and pharmacokinetics of AAPB for injection in healthy Chinese subjects.

The objective of this study was to evaluate the safety, tolerability, and pharmacokinetic characteristics of single and multiple intravenous infusion of AAPB at different doses for 7 consecutive days, and to explore the metabolites and mass balance of AAPB for injection in vivo. It provides a research basis for exploring the efficacy and safety of AAPB for injection in the treatment of acute ischemic death.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, aged between 18 and 45 (both ends included), both male and female;
2. When screening patients, male weight ≥50kg, female weight ≥45kg, body mass index (BMI) in the range of 19-28 kg/m^2 (including the upper and lower limits), BMI= weight (kg)/height (m) ^2;
3. Able to communicate well with researchers, willing and able to comply with the lifestyle restrictions specified in the program;
4. Women or men of reproductive age who agree to use investigatorial-approved contraceptive methods (such as Iuds, condoms, spermicide gel plus condoms, diaphragms, etc.) throughout the trial period;
5. Fully understand the purpose and requirements of the trial, voluntarily participate in the clinical trial and sign a written informed consent, and be able to complete the whole process of the trial according to the requirements of the trial.

Exclusion Criteria:

1. The investigator determines that the subject has a history of present disease and past disease or dysfunction affecting the clinical trial, including but not limited to diseases of the nervous system, cardiovascular system, respiratory system, digestive system, urinary system, endocrine system, metabolic disease, rheumatic disease, blood system, etc.;
2. Suffers from mental illness or has a history of mental illness;
3. Have a history of malignant tumors or other diseases that are not suitable for clinical trials;
4. History of cardiovascular disease (such as heart dysfunction, coronary artery disease, cardiomyopathy, valvular heart disease, family history of congenital long QT syndrome, family history of sudden death, etc.) or ECG results showing QTcF > 450ms, or clinically significant conduction block or T wave changes;
5. Abnormal liver function (ALT, AST higher than the upper limit of normal reference value);
6. Any drugs that inhibit or induce liver drug metabolism enzymes (such as: inducers barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole, etc.) were used within 30 days before drug administration; Inhibitors 5-hydroxyserotonin reuptake inhibitor (SSRI) antidepressants, cimetidine, Diltiazem, macrolides, nitroimidazoles, sedatives and hypnotics, verapamil, fluoroquinolones, antihistamines, etc. Or any prescription, over-the-counter, and herbal medicines other than those described above have been taken in the 14 days prior to drug administration;
7. Participated in any clinical trials within 3 months before enrollment;
8. Those who have special requirements for food and cannot comply with a unified diet;
9. People who consumed any caffeine-rich food or drink (coffee, tea, cola, chocolate, etc.) within 48 hours before the study drug administration, or who do not agree to prohibit the use of any caffeine-rich food or drink during the study period;
10. Known allergic history of test drug ingredients or similar drugs, allergic disease history or allergic constitution;
11. Smokers who smoked more than 10 cigarettes or equivalent cigarettes per day in the 1 year prior to screening, or those who could not comply with the prohibition of smoking during the test period;
12. Alcohol-addicted persons with an average weekly alcohol intake of more than 14 units (1 unit =285ml beer or 25ml spirits or 150ml wine) or positive for alcohol breath test in the year before screening;
13. Persons with a history of drug or drug abuse within the year prior to screening, or who test positive for drug abuse (screening items include: morphine, THC, methamphetamine, dimethylene dioxyamphetamine, ketamine and cocaine);
14. Complete physical examination, vital signs, laboratory examination, ECG examination determined by the investigator to be abnormal and clinically significant;
15. Hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), HIV antibody (HIV-AB), Treponema pallidum antibody (TP-Ab) any of the positive results;
16. Women who are pregnant or nursing, or who test positive for serum HCG before trial administration, or who are unable or unwilling to use investigator-approved contraception during the study period and for 3 months after the end of the study as directed by the investigator;
17. Study blood donation or blood loss ≥200ml within 3 months before drug administration, or have a history of blood product use;
18. Patients with a history of surgery within 3 months prior to study administration, or who have not recovered from surgery, or who have an anticipated surgical plan during the trial period;
19. Persons directly related to the clinical trial;
20. Patients who cannot tolerate venipunction and have a history of fainting needles and fainting blood;
21. Other subjects deemed unsuitable for this study by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-11-14 (Estimated); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Adverse event | Simple ascending dose, follow-up visit from day 1 to day 3. Multiple Ascending Dose, follow-up visit from day 1 to day 8.
  Incidence of Adverse Events

SECONDARY OUTCOMES:
Serum Human chorionic gonadotropin in female subjects of reproductive age | Screening period (day-14 ~ day-1)，Baseline Period (day0)，Final follow-up period(day3/day8)
Maximum plasma concentration (Cmax) | Day1~day2
  Blood will be drawn from adult subjects pre-drug application(within 60min) and at 30min, 60min, 90min, 120min, 180min, 240min (4h), 480min (8h），720min (12h)，1440min(24h).
Time to maximum plasma concentration (Tmax) | Day1-day2
  Blood will be drawn from adult subjects pre-drug application(within 60min) and at 30min, 60min, 90min, 120min, 180min, 240min (4h), 480min (8h），720min (12h)，1440min(24h).
Elimination half-life (t1/2) | Day1-day2
  Blood will be drawn from adult subjects pre-drug application(within 60min) and at 30min, 60min, 90min, 120min, 180min, 240min (4h), 480min (8h），720min (12h)，1440min(24h).
clearance, CL | Day1-day2
  Blood will be drawn from adult subjects pre-drug application(within 60min) and at 30min, 60min, 90min, 120min, 180min, 240min (4h), 480min (8h），720min (12h)，1440min(24h).
Apparent distribution volume (Vz) | Day1-day2
  Blood will be drawn from adult subjects pre-drug application(within 60min) and at 30min, 60min, 90min, 120min, 180min, 240min (4h), 480min (8h），720min (12h)，1440min(24h).
Steady statetime time to maximum plasma concentration （Tmax_ss） | Day1-day2， Day4-day8
  Day1，blood will be drawn from adult subjects pre-drug application(within 60min) and at 30min, 60min, 80min, 100min, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h .
  Day4，5，6，7，blood will be drawn from adult subjects pre-drug application(within 15 min) .
  Day7, blood will be drawn from adult subjects pre-drug application 30min, 60min, 80min, 100min, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h and 24h after administration.
steady state minimal concentration（Cmin,ss） | Day1-day2， Day4-day8
  Day1，blood will be drawn from adult subjects pre-drug application(within 60min) and at 30min, 60min, 80min, 100min, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h .
  Day4，5，6，7，blood will be drawn from adult subjects pre-drug application(within 15 min) .
  Day7, blood will be drawn from adult subjects pre-drug application 30min, 60min, 80min, 100min, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h and 24h after administration.
steady state maximum concentration（Cmax,ss） | Day1-day2， Day4-day8
  Day1，blood will be drawn from adult subjects pre-drug application(within 60min) and at 30min, 60min, 80min, 100min, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h .
  Day4，5，6，7，blood will be drawn from adult subjects pre-drug application(within 15 min) .
  Day7, blood will be drawn from adult subjects pre-drug application 30min, 60min, 80min, 100min, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h and 24h after administration.
Fluctuation Factor （DF） | Day1-day2， Day4-day8
  Day1，blood will be drawn from adult subjects pre-drug application(within 60min) and at 30min, 60min, 80min, 100min, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h .
  Day4，5，6，7，blood will be drawn from adult subjects pre-drug application(within 15 min) .
  Day7, blood will be drawn from adult subjects pre-drug application 30min, 60min, 80min, 100min, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h and 24h after administration.
steady state clearance（CLss） | Day1-day2， Day4-day8
  Day1，blood will be drawn from adult subjects pre-drug application(within 60min) and at 30min, 60min, 80min, 100min, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h .
  Day4，5，6，7，blood will be drawn from adult subjects pre-drug application(within 15 min) .
  Day7, blood will be drawn from adult subjects pre-drug application 30min, 60min, 80min, 100min, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h and 24h after administration.
12-lead electrocardiogram interpretation | Screening period (day-14 ~ day-1)，Baseline Period (day0)，Administration observation period (day1~3 /day1~8)， Final follow-up period(day3/day8)
  Heart Rate，Cardiac rhythm， ECG RR interval，ECG QRS Interval， ECG PR Interval，ECG QTcF Interval，
Blood pressure | Screening period (day-14 ~ day-1)，Baseline Period (day0)，Administration observation period (day1~3 /day1~8)， Final follow-up period(day3/day8)
  Blood pressure is recorded in millimeters of mercury
Respiration | Screening period (day-14 ~ day-1)，Baseline Period (day0)，Administration observation period (day1~3 /day1~8)， Final follow-up period(day3/day8)
  The unit of recording is the number of breaths per minute.
Heart rate | Screening period (day-14 ~ day-1)，Baseline Period (day0)，Administration observation period (day1~3 /day1~8)， Final follow-up period(day3/day8)
  The unit of heart rate is the number of heartbeats per minute.
Temperature | Screening period (day-14 ~ day-1)，Baseline Period (day0)，Administration observation period (day1~3 /day1~8)， Final follow-up period(day3/day8)
  Body temperature is recorded in degrees Celsius

CONTACTS AND LOCATIONS:
Overall Officials: Li shuya Director of Clinical Trial Center, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China